CLINICAL TRIAL: NCT03273231
Title: The Effect of Ketamine on Immune Function and Prognosis in Patients Undergoing Colorectal Cancer Resection
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 4-2017-0475
Record Dates: First submitted 2017-09-04; First posted 2017-09-06 (Actual); Last update posted 2019-01-16 (Actual); Status verified 2019-01

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Ketamine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ketamine group (Experimental): Ketamine is administered intravenously with a loading dose of 0.25 mg/kg at 5 minutes before surgery, followed by an infusion rate of 0.05 mg/kg/h to the end of surgery.
  Interventions: Drug: Ketamine
- control group (Placebo Comparator): 0.9% saline solution
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Ketamine — Ketamine is administered intravenously with a loading dose of 0.25 mg/kg at 5 minutes before surgery, followed by an infusion rate of 0.05 mg/kg/h to the end of surgery.
  Arms: ketamine group
Drug: Saline — 0.9% saline solution
  Arms: control group

SUMMARY:
Systemic inflammation caused by surgery may aggravate immunosuppression in immunocompromised cancer patients. The natural killer (NK) cell is a critical part of anti-tumor immunity. ketamine, a N-methyl-D-asparate receptor antangonist, has anti-inflammatory activity and opioid-sparing effect. This study investigate the effect of intraopertaive ketamine administration on immune function in patients undergoing laparoscopic colorectal cancer resection.

ELIGIBILITY:
Inclusion Criteria:

* patient between 20 and 80 of age with ASA physical status Ⅰ-Ⅲ
* patient scheduled for laparoscopic colorectal cancer resection

Exclusion Criteria:

* ASA physical status Ⅳ
* severe hepatorenal disease
* heart failure
* infection
* increased intracranial pressure, seizure
* preoperative chemotherapy
* immune or endocrine disease
* metastasis to other organ
* problem with communication
* pregnancy
* body mass index > 35 kg/m2

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-09-01 (Actual); Primary Completion 2020-07 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
natural killer cell cytotoxicity | Baseline
  Natural killer cell cytotoxicity is measured with NK Vue Kit™(ATGen, Gyeonggi-do, Korea).
natural killer cell cytotoxicity | 1 hour after surgery
  Natural killer cell cytotoxicity is measured with NK Vue Kit™(ATGen, Gyeonggi-do, Korea).
natural killer cell cytotoxicity | postoperative day 1
  Natural killer cell cytotoxicity is measured with NK Vue Kit™(ATGen, Gyeonggi-do, Korea).
natural killer cell cytotoxicity | postoperative day 2
  Natural killer cell cytotoxicity is measured with NK Vue Kit™(ATGen, Gyeonggi-do, Korea).

SECONDARY OUTCOMES:
proinflammatory cytokine | Baseline
  Inflammtory response is assesssed by measuring levels of proinflammtory cytokines.
proinflammatory cytokine | 1 hour after surgery
  Inflammtory response is assesssed by measuring levels of proinflammtory cytokines.
proinflammatory cytokine | postoperative day 1
  Inflammtory response is assesssed by measuring levels of proinflammtory cytokines.
proinflammatory cytokine | postoperative day 2
  Inflammtory response is assesssed by measuring levels of proinflammtory cytokines.
recurrence | 1 year after surgery
  Cancer recurrence is evaluated 1 year after surgery.
metastasis | 1 year after surgery
  Cancer metastasis is evaluated 1 year after surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine, Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cho JS, Kim NY, Shim JK, Jun JH, Lee S, Kwak YL. The immunomodulatory effect of ketamine in colorectal cancer surgery: a randomized-controlled trial. Can J Anaesth. 2021 May;68(5):683-692. doi: 10.1007/s12630-021-01925-3. Epub 2021 Feb 2. PMID 33532995